CLINICAL TRIAL: NCT05405153
Title: Urdu Version of Parkinson's Disease Questionnaire-8. A Cross-cultural Validity and Reliability Study
Brief Title: Translation of Parkinson's Disease Questionnaire -8 in Urdu Language
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Nayab Khurram
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: PDQ-8, Parkinson's disease, validate .
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross cultural analytical study to translate Parkinson's disease questionnaire-8 in Urdu language. Along with the translated version by evaluating its validity and reliability among the patients of Parkinson's disease. No such study has been previously conducted in Pakistan which translate this questionnaire in

Urdu and follows the proper cross- culture adaptation. Condition or disease:

Parkinson's disease. Convenient sampling technique would be used

DETAILED DESCRIPTION:
Parkinson's Disease Questionnaire-8 (PDQ-8) is the brief version of PDQ-39 formulated to reduce the respondent burden and for convenient use in clinical settings in patients of Parkinson's disease. (PDQ-8) is the patient reported outcome measure constructed by taking one question from each of the eight domains of PDQ-39 (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. PDQ-8 will be translated into Urdu language by Beaton et al guidelines for cross cultural adaptation of tool. The validity and reliability of Urdu version of PDQ-8 will be evaluated by calculating Cronbach's alpha, intra-class correlation coefficient and Pearson/spearman rank correlation co-efficient.

Continuous variables will be shown by mean and standard deviation and the categories will be demonstrated in frequency and percentage. Factor structure of the PDQ-8 will be extracted using exploratory factor analysis (EFA), utilizing principal component analysis with varimax rotation.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Both genders
* Patients with diagnosed Idiopathic Parkinson's disease (IPD) by neurophysician
* Patient able to read Urdu Language. Patients who can participate in community, patients with cognitive issue, Patients with MMSE more than 24 will be included

Exclusion Criteria:

* Patients with any other neurological issue
* Patients who undergo brain surgery

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Parkinson's disease questionnaire (PDQ-8) | 8 months
  Parkinson's disease Questionnaire-8 (PDQ-8) is the brief version of PDQ-39 formulated to reduce the respondent burden and for convenient use in clinical settings in patients of Parkinson's disease. (PDQ-8) is the patient reported outcome measure constructed by taking one question from each of the eight domains of PDQ- 39 (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort)

SECONDARY OUTCOMES:
Reliability of translated versions of PDQ-8 | 8 months
  To determine the reliability of cross-culturally adapted and translated PDQ-8 in the patients with Parkinson's disease. Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two intervals between different visits of the patient. Thus, the reliability of tool will be assessed by internal consistency and test-retest reliability
Validity of translated versions of PDQ-8 | 8 months
  To determine the validity of cross-culturally adapted and translated PDQ-8 in the patients with Parkinson's disease.
  Validity is how accurate the results are.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhan A, Mohan S, Tarolli C, Schneider RB, Adams JL, Sharma S, Elson MJ, Spear KL, Glidden AM, Little MA, Terzis A, Dorsey ER, Saria S. Using Smartphones and Machine Learning to Quantify Parkinson Disease Severity: The Mobile Parkinson Disease Score. JAMA Neurol. 2018 Jul 1;75(7):876-880. doi: 10.1001/jamaneurol.2018.0809. PMID 29582075
- [Background] Ellis TD, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Thackeray A, Thiese MS, Dibble LE. Identifying clinical measures that most accurately reflect the progression of disability in Parkinson disease. Parkinsonism Relat Disord. 2016 Apr;25:65-71. doi: 10.1016/j.parkreldis.2016.02.006. Epub 2016 Feb 2. PMID 26876037